CLINICAL TRIAL: NCT00775320
Title: Assessment of Suspected Intracranial Malignancy Using 3'-Deoxy-3'18 F-fluorothymidine Positron Emission Tomography
Brief Title: Assessment of Suspected Intracranial Malignancy Using 3'-Deoxy-3'18 F-flourothymidine PET
Status: Terminated | Type: Observational
Why Stopped: Study closed by institutional review board
Sponsor: University of Oklahoma (Other)
Collaborators: Midwest Medical Isotopes (Unknown)
Responsible Party: Sponsor
Other Study IDs: FLT- Brain Study
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Brain Tumor
Keywords: Brain scan
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue from brain tumor
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Brain tumor FLT-PET: Those diagnosed with a brain tumor and are to undergo surgery
  Interventions: Procedure: FLT-PET scan

INTERVENTIONS:
Procedure: FLT-PET scan — Imaging test

SUMMARY:
The primary objective of this study is to detect and quantify tumor cells of high grade malignant gliomas and metastatic brain lesions both before and after initial surgical resection in a cohort of newly diagnosed patients.

DETAILED DESCRIPTION:
In this study, 35 patients will be selected to undergoing sequential imaging with FLT-PET. Prior to surgical resection, patients will undergo a preliminary FLT-PET. Additional FLT scans for a maximum of four scans.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Women must not be pregnant or breast feeding
* Histologic or strong radiologic suspicion of high grade malignant glioma or ogliometastatic tumor(s)

Exclusion Criteria:

* May not have received previous therapy for their malignancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with a brain tumor and to undergo surgery
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2008-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Holter, MD, Principal Investigator — Assistant Professor
Locations (1):
- University Of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States